CLINICAL TRIAL: NCT04872829
Title: Comparative Analysis of Visual Outcomes of Multifocal and Monofocal Intraocular Lenses in Congenital Cataract Surgery
Brief Title: Multifocal vs Monofocal IOL in Congenital Cataract Surgery
Status: Completed | Type: Observational
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Luca Buzzonetti, Head of the Ofthalmology Departement, Bambino Gesù Hospital and Research Institute
Other Study IDs: L121
Record Dates: First submitted 2021-04-26; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Cataract Congenital
MeSH Terms: interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- multifocal IOL group: patients with unilateral and bilateral multifocal IOL
  Interventions: Device: cataract surgery
- monofocal IOL group: patients with unilateral and bilateral monofocal IOL
  Interventions: Device: cataract surgery

INTERVENTIONS:
Device: cataract surgery — All patients underwent cataract surgery under 1 year of age (mean age 8 months, range 6-12) performed with the same surgical technique: two 1.2 mm clear corneal incision, continuous curvilinear capsulorhexis with a diameter of approximately 6.0 mm and intraocular lens implantation, posterior capsulotomy and anterior vitrectomy.
  IOL power was calculated using Sanders-Retzlaff-Kraff (SRK)/II formula. Multifocal IOL implantated was Alcon AcrySof ReSTOR SN60D3, while the monofocal one was Alcon AcrySof SN60AT.
  According to the Infant Aphakia treatment Study, the IOL power was calculated as a function of the child age17, with an undercorrection ranging from 4 to 6 D.

SUMMARY:
The aim of this study is to evaluate long-term outcome after congenital cataract surgery comparing results achieved with multifocal and monofocal IOLs.

DETAILED DESCRIPTION:
PURPOSE: To assess the impact on visual development of multifocal versus monofocal intraocular lenses (IOLs) implantation in children following congenital cataract surgery.

DESIGN: Retrospective interventional consecutive case series. METHODS: We reviewed the records of 56 eyes of 43 pediatric patients who underwent congenital cataract surgery with phacoaspiration and simultaneous implantation of IOL under one year of age. Corrected distance visual acuity (CDVA), refractive error and ocular motility disorders were evaluated after a follow-up greater than 4 years.

ELIGIBILITY:
Inclusion Criteria:

* unilateral congenital cataract
* bilateral congenital cataract

Exclusion Criteria:

* other ocular pathologies (such as glaucoma, microphthalmia, micro - or megalocornea, persistent fetal vasculature, retinal congenital disease, corneal scar, traumatic cataracts)
* systemic diseases (such as chromosomal abnormalities, prematurity or mental retardation)

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We reviewed the records of 56 eyes of 43 pediatric patients who underwent congenital cataract surgery with phacoaspiration and simultaneous implantation of IOL under one year of age. All patients were directed to our hospital from primary care ophthalmologists or pediatricians
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2008-06-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Mean CDVA | CDVA was evaluated after 4 years of age.
  Corrected distance visual acuity (CDVA), calculated in logarithm of the minimum angle of resolution (logMAR), using standard Snellen charts

CONTACTS AND LOCATIONS:
Overall Officials: Luca Buzzonetti, MD, Principal Investigator — Bambino Gesù Children's Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: No
All the data are stored in the Bambino Gesù Children's Hospital data base

REFERENCES:
- [Derived] Buzzonetti L, Petroni S, De Sanctis CM, Valente P, Federici M, Benassi C, Iarossi G. Comparative analysis of visual outcomes of multifocal and monofocal intraocular lenses in congenital cataract surgery. J Cataract Refract Surg. 2022 Jan 1;48(1):56-60. doi: 10.1097/j.jcrs.0000000000000705. PMID 34054076